CLINICAL TRIAL: NCT02621008
Title: A Self-Administered Mobile Phone-based Holistic Intervention for Promoting Healthy Habits and Weight Loss in People Who Are Overweight or Obese
Brief Title: Mobile Phone-based Intervention for Promoting Healthy Habits and Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eco Fusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Hypertension; Pre-diabetes; Overweight; Obese; Weight; Adherence
Keywords: diabetes; hypertension; obesity; mobile phone; stress; healthy living; pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Glucose Intolerance; Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress Reduction& Healthy living (Experimental): Utilizing a stress reduction app (Serenita) and lifestyle intervention App (NewMe) and obtaining the NewMe guideline for healthy living, plus obtaining periodic messages regarding healthy living.
  Interventions: Other: Stress Reduction& Healthy living

INTERVENTIONS:
Other: Stress Reduction& Healthy living — Utilizing a stress reduction app (Serenita) and lifestyle intervention App (NewMe) and obtaining the NewMe guideline for healthy living, plus obtaining periodic messages regarding healthy living.

SUMMARY:
A self administered 16 weeks plus follow up study to explore the efficacy of mobile phone driven apps for stress reduction coupled with guidance for healthy living among obese and overweight populations. The Study primary end points are weight of the participants, as well as glucose measurements (for subject with diabetes) and blood pressure (of subjects with hypertension).

DETAILED DESCRIPTION:
The NewMe™ (Eco-fusion, Ltd) is a science driven lifestyle change program for better living (www.eco-fusion.com).

What's in the program? It starts with two weeks to shakeup the patient. It is focused on ridding the patient of known food addictions and helping the body patient return to its long forgotten normal operating environment. The patient is expected to notice a dramatic change in its well-being after those two weeks.

The NewMe program uses mobile health and motivational psychology to help impact sustainable lifestyle changes. The program takes a holistic approach to the etiology of adverse lifestyle habits and personalizes the solution to each individual. It is based on a variety of clinical constructs, including multiple studies related to biofeedback and stress relief, appended with the latest scientific development in nutrition and fitness, and enhanced with a technology platform specifically developed to deliver such care. The goal of the program is rapid and sustainable life changes with measurable parameters such as increased quality of life, reduced stress level, improved blood pressure and cholesterol, blood sugar and weight.

At the core of the system is a comprehensive clinical program combining nutrition, stress management, fitness, and social support, guided by a suite of software apps and emails which guide participants through a 16 weeks program, which is kick-started by a 2 weeks Rapid Start up Regimen. The solution combines a structured program and interactions and teaches participants how to integrate a healthier routine into their day-to-day life.

Core content include a broad behavioral focus on the principles of making healthy food choices and meal planning, instructions on how to combine both healthy diet and inclusion of an activity, stress & sleep tracker. Stress gets special attention with the integration of breathing exercises, biofeedback training & meditation into a daily routine in order to control and reduce emotional eating and other eating binges. This is done through the Serenita App.

To promote behavior change, the program introduces the cognitive and behavioral strategies, critical for long-term disease reversal. Other instructional content relates to the importance of including a modified high-nutrient density and fiber, low- caloric density foods in meal planning (although there is no caloric restriction in the program), managing self-defeating thinking patterns, and incorporating both fat burning & strength training into a physical activity regime.

The program is divided into 2 stages:

* Stage One - Week 1 & 2- Rapid Start up regimen, in which the participants follow a nutrient rich, low processed and carbs dietary regimen.
* In addition, using a personalized sensor driven app, participants practice daily breathing exercises & guided meditation, intended to manage stress, and control food cravings. Physical activity regimen is also integrated into the daily routine. They confirm and log their daily activity which is software guided
* Stage two, weeks 3-16. During this period some of the restricted foods in Stage one are being reintroduced and the effect of reintroduction is explored.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older and
* have a body mass index (BMI) of at least 24 kg/m2 (22 kg/m2 if Asian) and
* be able to engage in light physical activity

Exclusion Criteria:

* no Internet access or use of iOS
* taking more than three antihypertensive or diabetes drugs; meeting the DSM-5 criteria for an eating disorder
* having a disability that prevents or hinders exercise and physical activity
* receiving any treatment for weight loss elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
BMI | 16 weeks
Glucose level | 16 weeks
blood pressure | 16 weeks
BMI | 6 months
BMI | 12 months
glucose level | 6 months
glucose level | 12 months
blood pressure | 6 months
blood pressure | 12 months

SECONDARY OUTCOMES:
Quality of Life questionnaire | 16 weeks
Quality of Life questionnaire | 6 months
Quality of Life questionnaire | 12 months
Burnout measure | 16 weeks
Burnout Measure | 6 months
Burnout measure | 12 months
Perceived dietary adherence questionnaire | 16 weeks
Perceived dietary adherence questionnaire | 6 months
Perceived dietary adherence questionnaire | 12 months
Mind wandering index | 16 weeks
  tendency and frequency of mind wandering
Mind wandering index | 6 months
Mind wandering index | 1 year
stress mindset scale | 16 weeks
stress mindset scale | 6 months
stress mindset scale | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mt Sinai Medical Center, New York, New York, United States